CLINICAL TRIAL: NCT04411134
Title: A Phase I Study of E7 TCR T Cell Immunotherapy for High-Grade Cervical Intraepithelial Neoplasia
Brief Title: E7 TCR T Cell Immunotherapy for High-Grade Cervical Intraepithelial Neoplasia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed based on the lack of perceived clinical activity observed from a different study treating a similar patient population with same study agent.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200093; 20-C-0093
Record Dates: First submitted 2020-05-30; First posted 2020-06-02 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: T Cell Receptor; Immunotherapy; Human Papillomavirus; Intralesional Injections; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Approximately 3x10^8 or 1.5x10^9 E7 TCR T cells will be injected on day 0 and 1.5x10^9 E7 TCR T cells on day 31 (2 escalating dose levels)
  Interventions: Biological: E7 TCR
- Arm 2 (Experimental): The MTD from among dose level 1 and dose level 2
  Interventions: Biological: E7 TCR

INTERVENTIONS:
Biological: E7 TCR — Approximately 3x10^8 or 1.5x10^9 E7 TCR T cells will be injected on day 0 and 1.5x10^9 E7 TCR T cells on day 31 (2 escalating dose levels)

SUMMARY:
Background:

Human papillomavirus (HPV) can lead to High-Grade Cervical Intraepithelial Neoplasia (CIN 2,3). This type of lesion has a high risk of becoming cancer. T cells are part of the immune system. A new type of treatment involves modifying these cells and injecting them into the lesions to shrink them.

Objective:

To test if injecting a type of treatment directly into cervical lesions can be safely given as therapy for high-grade CIN.

Eligibility:

People ages 21 and older with CIN 2,3 caused by HPV-16

Design:

Participants will be screened over at least 2 visits with:

Tumor sample

Blood and urine tests

Medical and medication history

Physical exam

Pelvic exam and colposcopy to look at the cervix

Participants will have a baseline visit. They may be admitted to the hospital. They may receive a large catheter inserted into a vein. They will have a vein assessment.

Before they receive treatment, participants will have a biopsy of the cervix. They will have leukapheresis. Blood will be removed through a needle in the arm, circulated through a machine that takes out the while blood cells, then returned through a needle in the other arm. A central catheter may also be used.

Participants will have the modified cells injected directly into their cervical lesions. They will recover in the hospital for 1-2 days.

Participants will have follow-up visits 2 weeks, 31 days, 6 weeks, and 12 weeks after treatment. They may receive a second injection at the 31-day visit.

Participants will be contacted once a year for 5 years after treatment. They will be followed for up to 15 years.

DETAILED DESCRIPTION:
Background:

* Cervical Intraepithelial Neoplasia (CIN) is caused by persistent infection with the Human Papillomavirus (HPV).
* High-grade lesions are common, affecting 5% of the female population in the United States, and are more likely to progress to cervical cancer.
* Surgical and ablative therapies are effective but can lead to long-term morbidity. New treatment modalities are needed.
* E7 TCR T cells have demonstrated safety and clinical activity in treatment-refractory metastatic HPV+ cancers.

Objectives:

- To determine the safety of intralesional injection of E7 TCR T cells as therapy for high- grade CIN.

Eligibility:

- Patients greater than or equal to 21 years of age with HPV16-associated, high-grade CIN.

Design:

* This is a phase I clinical trial with a 3+3 dose escalation design.
* Patients will receive intralesional injections of E7 TCR T cells.
* Patients will not receive a conditioning chemotherapy regimen or systemic aldesleukin.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed high-grade cervical intraepithelial neoplasia (CIN 2,3). Confirmation of high-grade cervical intraepithelial neoplasia (pathology report from outside institution is sufficient). Pathology confirming high-grade CIN must be within 3 months prior to initiation of study therapy. If needed, confirmatory biopsy of lesion(s) may be performed.
* HPV16+ CIN 2,3 and HLA-A*02:01 HLA type
* Patients may be treatment-naive or have received previous treatment for high-grade CIN. Patients who have received previous treatment are eligible if prior treatment was greater than or equal to 3 months before first dose of E7 TCR T cells and there is pathological confirmation of recurrent or persistent disease. If needed, confirmatory biopsy of lesion(s) may be performed.
* Patients can have either one lesion or multiple lesions with at least one lesion being visible on colposcopy to help facilitate intralesional administration of E7 TCR T cells.
* Age greater than or equal to 21 years. Because treatment for this disease is not recommended in patients <21 years of age, children and adolescents <21 years old are excluded from this study.
* ECOG performance status greater than or equal to 2.
* Patients must have adequate organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin within 1.5X normal institutional limits
  * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits
  * creatinine clearance Calculated creatinine clearance (CrCl) >50mL/min/1.73m^2 for patient with creatinine levels above institutional normal (by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation)
* Women of child-bearing potential must have a negative pregnancy test because E7 TCR T cells have unknown potential for teratogenic or abortifacient effects. Women of childbearing potential are defined as all women who are not post-menopausal or who have not had a hysterectomy. Postmenopausal will be defined as women over the age of 55 who have not had a menstrual period in at least 1 year.
* The effects of E7 TCR T cells on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (intrauterine device, hormonal or barrier method of birth control, abstinence, tubal ligation or vasectomy) prior to study entry and for up to 4 months after treatment. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
* Seronegative for HIV antibody. The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment.
* Seronegative for hepatitis B antigen and hepatitis C antibody. If hepatitis C antibody test is positive, then the patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Must be willing to participate in Gene Therapy Long Term Follow up Protocol, which will follow patients for up to 15 years per Food and Drug Administration (FDA) requirements.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with E7 TCR T cells, breastfeeding should be discontinued if the mother is treated with E7 TCR T cells. These potential risks may also apply to other agents used in this study.
* Patients with any form of systemic immunodeficiency, including acquired deficiency such as HIV or primary immunodeficiency such as Severe Combined Immunodeficiency Disease, are ineligible. The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the treatment.
* Patients on immunosuppressive drugs including systemic corticosteroids (inhaled or intranasal corticosteroids are allowed).
* Patients with a second active invasive cancer are not eligible.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
To determine the safety of intralesional injection of E7 TCR T cell therapy for highgrade CIN | 3 months
  The fraction who experience a DLT based on the dose level and cell administration within the dose level will be determined and reported.The analysis will be entirely descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Hinrichs, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0093.html